CLINICAL TRIAL: NCT06217783
Title: Ultrasound-guided Peripheral Intravenous Catheter Placement in an Oncologic Emergency Department - a Prospective, Randomized Controlled Trial of Catheter Lengths
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023-0848; NCI-2024-00503 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-01-10; First posted 2024-01-22 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Oncologic Complications and Emergencies
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Group A (Experimental): Participants will receive a catheter that is up to 1.75 inches long based on what the nurse thinks is best for you.
  Interventions: Device: Introcan Safety IV Catheter
- Group B (Experimental): Participants will receive a catheter that is either 1.75 or 2.5 inches long based on what the nurse thinks is best for you.
  Interventions: Device: Introcan Safety IV Catheter

INTERVENTIONS:
Device: Introcan Safety IV Catheter — Given by IV

SUMMARY:
To learn about the effects of the length of the catheter on the failure and success rate of USIV placement.

DETAILED DESCRIPTION:
Primary Objectives:

- The rate of catheter failure, defined as removal of the catheter for any reason other than "Care Complete" (i.e. a composite of removal due to "infiltration," "leaking," "catheter damage," "occlusion"), by day 10.

Secondary Objectives:

1. Time from catheter placement to removal (i.e. survival or dwell time).
2. Per catheter length rate of failure analysis
3. Rate of repeat catheterization
4. Rate of infection
5. Rate of thrombosis

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old.
2. Provision of signed and dated informed consent form.
3. Predetermined to have difficult IV access necessitating USIV placement
4. Expected admission to hospital with anticipated stay > 48 hours (per discussion with treating physician).

Exclusion Criteria:

1. Expected/anticipated discharge disposition from the ACCC (per discussion with treating physician).
2. Inability to give informed consent.
3. Pregnant women.
4. Non-English speaking participants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-03-27 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Rowland, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org